CLINICAL TRIAL: NCT02188641
Title: EFFECT OF EXERCISE AND DIETARY WEIGHT LOSS ON SYMPTOMS AND SYSTEMIC INFLAMMATION IN OBESE ADULTS WITH PSORIATIC ARTHRITIS: RANDOMIZED CONTROLLED TRIAL
Brief Title: Effect of Exercise and Diet on Psoriatic Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alexandria (Other)
Responsible Party: Principal Investigator, Anna Abou-Raya, MD, University of Alexandria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: alexmed12671300
Record Dates: First submitted 2014-07-04; First posted 2014-07-11 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2014-07

CONDITIONS: Psoriatic Arthritis
Keywords: Psoriatic arthritis; inflammation; obesity; diet; exercise
MeSH Terms: conditions — Arthritis, Psoriatic; Inflammation; Obesity; Motor Activity | interventions — Diet; Exercise; Population Groups

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Diet (Other): Low-fat diet
  Interventions: Other: Diet
- Exercise (Other): 3-day/week exercise programme
  Interventions: Other: Exercise
- Diet and exercise (Other): healthy low fat diet and 3day/week exercise programme
  Interventions: Other: Diet and Exercise
- Healthy lifestyle (Control) group (Other): Control group was provided with health education using videotaped presentation
  Interventions: Other: Healthy Lifestyle (Control) Group

INTERVENTIONS:
Other: Diet
  Arms: Diet
Other: Exercise
  Arms: Exercise
Other: Diet and Exercise
  Arms: Diet and exercise
Other: Healthy Lifestyle (Control) Group
  Arms: Healthy lifestyle (Control) group

SUMMARY:
Psoriatic arthritis (PsA) is a particular pattern of inflammatory arthritis often seen in association with psoriasis. PsA patients have a higher prevalence of comorbidities including obesity, metabolic syndrome, depression and premature cardiovascular disease. There is evidence that obesity is associated with PsA. A 12 month study was conducted to determine whether exercise and dietary weight loss are more efficacious, either separately or in combination, than standard care alone in improving symptoms and signs in obese adults with PsA.

Fifty-five obese PsA patients with a body mass index (BMI) ≥30, were recruited. Patients were randomized into usual lifestyle (controls), diet only, exercise only, and diet plus exercise groups for 12 months. Disease activity was assessed. Blood samples collected after 12 hours overnight fasting were analysed for glucose, lipid profile, ESR, hsCRP, proinflammatory cytokines; tumour necrosis factor alpha (TNF-alpha), interleukin-6 (IL-6) and interleukin-17 (IL-17). The primary outcome measures included improvement in ACR20. Secondary endpoints included reduction in PASI score, DAS28-CRP response and physician and patient global assessment (PGA). Safety and tolerability were also assessed. Data was collected at baseline and every 6 months.

DETAILED DESCRIPTION:
There is evidence that obesity is associated with PsA. Obesity leads to increased proinflammatory cytokines which may contribute to the development of multiple disturbances in PsA patients.

A 12 month, randomized single blind clinical trial was conducted to determine whether long-term exercise and dietary weight loss are more efficacious, either separately or in combination, than standard care alone in improving physical function, pain, fatigue, depression and systemic inflammation in obese adults with PsA.

Fifty-five obese ethnically homogenous adult PsA patients with a body mass index (BMI) ≥30, who satisfied the classification of psoriatic arthritis criteria were recruited. Patients were randomized into usual lifestyle (controls), diet only, exercise only, and diet plus exercise groups together with the continued use of standard treatment.

Exclusion criteria included other inflammatory conditions. Detailed skin and rheumatological assessment was conducted. Disease activity was assessed by psoriasis area and severity index (PASI), disease activity score (DAS28CRP), Health Assessment Questionnaire- Disability Index (HAQ-DI), Beck's Depression Inventory (BDI) and fatigue numeric rating scale. Blood samples collected after 12 hours overnight fasting were analysed for glucose, lipid profile, ESR, hsCRP, proinflammatory cytokines; tumour necrosis factor alpha (TNF-alpha), interleukin-6 (IL-6) and interleukin-17 (IL-17). The primary outcome measures included improvement in ACR20, systemic inflammation markers, BMI, physical function, pain, fatigue, depression and HAQ-DI. Secondary endpoints included reduction in PASI score, DAS28-CRP response and physician and patient global assessment (PGA). Safety and tolerability were also assessed. Data was collected at baseline and every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* PsA patients with a body mass index (BMI) ≥30
* Must satisfy the classification of psoriatic arthritis criteria

Exclusion Criteria:

* Other inflammatory conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2013-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
ACR20 response | 12 months

SECONDARY OUTCOMES:
PASI score | 12 months
DAS28-CRP response | 12 months
physician global assessment (PGA) | 12 months
patient global assessment (PGA) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Anna Abou-Raya, MD, Principal Investigator — University of Alexandria
Locations (1):
- University of Alexandria, Alexandria, Alexandria Governorate, Egypt